CLINICAL TRIAL: NCT07326059
Title: An Observational Study on the Safety and Outcomes of MUSE Stem Cell Therapy in Participants With Traumatic Brain Injury Receiving International Clinical Treatment
Brief Title: Safety and Outcomes of MUSE Stem Cell Therapy in Individuals With Traumatic Brain Injury
Acronym: MUSE-TBI-OBS
Status: Not yet recruiting | Type: Observational
Sponsor: Healing Hope International (Other)
Responsible Party: Sponsor
Other Study IDs: HHI-TBI-MUSE-001
Record Dates: First submitted 2025-12-08; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Traumatic Brain Injury; Traumatic Brain Injury (TBI) Patients; Traumatic Brain Injury (TBI); Concussion, Initial Encounter; Traumatic Brain Injury (TBI); Concussion, Subsequent Encounter; Traumatic Brain Injury With Brief Loss of Consciousness; Traumatic Brain Injury With Persistent Cognitive Deficits
Keywords: MUSE Cells; Stem Cell Therapy; Regenerative Medicine; Traumatic Brain Injury; Chronic Brain Injury; Acquired Brain Injury; Cell-Based Therapy; Neuroregeneration; Adult Neurorehabilitation; Medical Tourism; Observational Study; Real-World Evidence; Healing Hope International; Functional Recovery; Compassionate Use Registry
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion; Brain Injury, Chronic; Brain Injuries

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MUSE Therapy Recipients With Chronic TBI: This cohort includes individuals aged 6 to 75 with chronic traumatic brain injury (TBI) who independently elect to receive MUSE (Multilineage-differentiating Stress-Enduring) stem cell therapy at licensed international treatment centers outside the United States. The study does not provide or administer the therapy; instead, it observes and documents real-world outcomes following treatment. Participants may receive MUSE cell infusions using varying doses, cell sources, and routes of administration, depending on the clinical site they choose. The study will collect longitudinal data on neurological function, quality of life, functional independence, and any adverse events over a 12-month follow-up period.
  Interventions: Biological: MUSE Stem Cell Therapy

INTERVENTIONS:
Biological: MUSE Stem Cell Therapy — MUSE (Multilineage-differentiating Stress-Enduring) stem cell therapy refers to the use of a naturally occurring subpopulation of mesenchymal lineage cells characterized by stress tolerance, expression of SSEA-3, and the capacity to differentiate into multiple cell types. Preclinical studies have shown that MUSE cells can migrate to sites of tissue injury, including the central nervous system, and may contribute to tissue repair through paracrine and regenerative mechanisms.
  In this observational study, participants independently obtain MUSE stem cell therapy at licensed treatment facilities outside the United States as part of their personal medical care. The study team does not provide, administer, manufacture, or direct the therapy.

SUMMARY:
This prospective observational study evaluates the safety profile and patient-reported outcomes associated with MUSE (Multilineage-differentiating Stress-Enduring) stem cell therapy in individuals aged 6 to 75 with chronic traumatic brain injury (TBI). Participants independently elect to receive MUSE cell treatment through international clinical programs, and this study aims to capture real-world evidence on the potential therapeutic effects and risks of this emerging regenerative approach.

The study does not administer any intervention. Instead, it follows participants who have received, or plan to receive, MUSE cell infusions outside the United States. Over a 12-month follow-up period, data will be collected on neurological functioning, quality of life, activities of daily living, and any reported adverse events or complications. Information will be gathered through remote interviews, structured digital surveys, and review of medical documentation when available.

This research is sponsored by Healing Hope International and is intended to contribute to the ethical and responsible advancement of novel cell-based therapies by generating real-world evidence that may guide future clinical trial development and inform patient care practices.

DETAILED DESCRIPTION:
This observational study is designed to systematically evaluate the safety, tolerability, and potential neurological outcomes associated with MUSE (Multilineage-differentiating Stress-Enduring) stem cell therapy in individuals with chronic traumatic brain injury (TBI) who independently obtain treatment through international clinical programs.

MUSE cells are a distinct subpopulation of mesenchymal stem cells characterized by stress resilience, spontaneous triploblastic differentiation, and the capacity to home to sites of tissue injury. Preclinical research suggests that MUSE cells may contribute to neuroregeneration through differentiation into neural and glial lineages, modulation of inflammatory pathways, and repair of damaged central nervous system structures. While early findings are promising, clinical evidence remains limited, highlighting the need for structured real-world data.

This study does not randomize participants or administer any treatment. Instead, it functions as a registry-style, real-world evidence platform following individuals who have elected to receive MUSE cell therapy at licensed facilities outside the United States. Collected data will include baseline demographics, TBI history, details of the stem cell procedure (such as cell source, administered dose, and route of delivery), and longitudinal follow-up over 12 months.

Primary domains of interest include:

Neurological function, assessed with validated clinical instruments (e.g., Glasgow Outcome Scale-Extended).

Quality of life, measured using standardized patient-reported outcome tools (e.g., PROMIS-29, EQ-5D).

Functional abilities and activities of daily living, to assess practical day-to-day impact.

Safety and tolerability, including documentation of adverse events, patient-reported symptoms, and any medical complications.

Data will be obtained through remote telemedicine visits, structured digital surveys, and review of available medical records. This study does not collect biospecimens and does not involve the administration of any investigational product.

The overarching objective is to generate high-quality real-world evidence regarding the use of MUSE stem cells in chronic TBI, supporting the scientific foundation needed for future controlled clinical trials and potential compassionate use pathways. The study is conducted by Healing Hope International, a nonprofit organization dedicated to advancing ethical access and research in regenerative medicine.

ELIGIBILITY:
Inclusion Criteria:

Individuals aged 6 to 75 years at the time of enrollment.

Documented history of traumatic brain injury (TBI) occurring at least 6 months prior to enrollment (chronic phase).

Participant has independently elected to receive MUSE (Multilineage-differentiating Stress-Enduring) stem cell therapy at a licensed treatment facility outside the United States.

Ability of the participant or legally authorized representative to provide informed consent for participation in an observational study.

Willingness to participate in remote or in-person follow-up assessments for up to 12 months.

Ability to provide medical records, laboratory reports, or treatment documentation when available.

Exclusion Criteria:

Individuals who have not received, and do not plan to receive, MUSE cell therapy as part of their independent medical care.

Inability or unwillingness to complete study assessments (e.g., severe communication barriers not manageable through caregiver assistance or technology).

Any condition that, in the opinion of the study team, would make participation in an observational registry unsafe or infeasible (e.g., inability to provide minimal required data).

Planned participation in another research study that would prevent collection of observational outcomes for this registry.

Individuals currently incarcerated or in institutional settings where research participation is restricted.

-

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study population consists of individuals aged 6 to 75 with chronic traumatic brain injury who independently choose to receive MUSE stem cell therapy at licensed medical facilities outside the United States. Participants represent a real-world cohort seeking regenerative treatment as part of their personal medical care. The study does not administer therapy but follows these individuals longitudinally to document safety signals, functional outcomes, quality-of-life measures, and health care utilization over a 12-month period. Data are collected through remote assessments, participant-provided medical documentation, and available clinical records.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2028-01 (Estimated); Primary Completion 2034-12 (Estimated); Study Completion 2036-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in global functional outcome (Glasgow Outcome Scale-Extended) | Baseline (pre-MUSE cell treatment) and 12 months after first MUSE cell treatment
  The Glasgow Outcome Scale-Extended (GOSE) is an 8-point ordinal scale (1 = Death, 8 = Upper Good Recovery) used to evaluate global functional status following traumatic brain injury. Higher scores reflect better functional outcome. This observational study will measure the change in GOSE score from baseline to 12 months after the participant's first independently obtained MUSE cell therapy session. Assessments will be conducted through structured interviews via in-person visits or telehealth, following standardized GOSE scoring procedures.

SECONDARY OUTCOMES:
Change in post-concussive symptoms (Rivermead Post-Concussion Symptoms Questionnaire) | Baseline; 3, 6, and 12 months after first MUSE cell treatment
  The Rivermead Post-Concussion Symptoms Questionnaire (RPQ) is a patient-reported outcome measure used to assess the severity of common post-concussive symptoms. The RPQ includes 16 items, each scored from 0 to 4, producing a total score range of 0-64, with higher scores indicating greater symptom severity. This study will evaluate the change in RPQ total score from baseline to each follow-up time point. Assessments will be conducted remotely using standardized RPQ administration procedures.
Change in cognitive function (Montreal Cognitive Assessment) | Baseline; 6 and 12 months after first MUSE cell treatment
  The Montreal Cognitive Assessment (MoCA) is a 30-point screening instrument used to evaluate global cognitive function across multiple domains, including attention, memory, executive functioning, language, and visuospatial abilities. Higher scores indicate better cognitive performance. This study will assess change in total MoCA score from baseline to 6- and 12-month follow-up visits. Assessments will be conducted using standardized MoCA administration procedures via in-person or telehealth formats.
Change in Health-Related Quality of Life Measured by EQ-5D-5L Index Score | Baseline; 6 and 12 months after first MUSE cell treatment
  Health related quality of life will be assessed using the EuroQol 5-Dimension 5-Level Questionnaire (EQ-5D-5L). The EQ-5D-5L measures health status across five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Responses are converted into a single summary health utility index score using country-specific value sets.
  Scale range: Typically less than 0 (health states worse than death) to 1.0 (perfect health)
  Interpretation: Higher EQ-5D-5L index scores indicate better overall health-related quality of life
  Changes in EQ-5D-5L index scores will be evaluated from baseline to follow-up assessments.
Change in functional independence (Functional Independence Measure) | Baseline; 6 and 12 months after first MUSE cell treatment
  Functional independence will be assessed using the Functional Independence Measure (FIM), an 18-item scale with total scores ranging from 18 to 126, higher scores indicating greater independence in activities of daily living. The outcome will be change in FIM total score from baseline to 6 and 12 months.
Change in mood and anxiety symptoms (HADS) | Baseline; 6 and 12 months after first MUSE cell treatment
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item self-report questionnaire with two subscales-HADS-Anxiety and HADS-Depression-each scored from 0 to 21, with higher scores indicating more severe symptoms. This study will evaluate changes in HADS-Anxiety and HADS-Depression subscale scores from baseline to 6- and 12-month follow-up assessments. The HADS will be administered using standardized procedures through remote or in-person data collection.
Change in Interleukin-6 (IL-6) Serum Concentration | Baseline; 3 and 6 months after first MUSE cell treatment
  Serum concentrations of Interleukin-6 (IL-6), a pro-inflammatory cytokine associated with chronic traumatic brain injury, will be obtained when available from participants' independently ordered clinical laboratory tests. IL-6 values will be abstracted from medical records or participant-provided laboratory reports. The study team does not order laboratory testing, collect biospecimens, or perform assays.
  Unit of measure: picograms per milliliter (pg/mL)
  Interpretation: Higher IL-6 concentrations indicate greater systemic inflammation
  Changes in IL-6 concentrations will be evaluated between baseline and follow-up time points.
Incidence of treatment-emergent serious adverse events | From first MUSE cell treatment through 12 months of follow-up
  Serious adverse events (SAEs) will be documented using participant reports and available medical records. SAEs will be classified according to ICH and FDA definitions, including events resulting in death, life-threatening conditions, hospitalization or its prolongation, persistent or significant disability/incapacity, or other medically significant events. This study will record the number and proportion of participants experiencing at least one SAE, as well as the total number of SAEs reported during the observation period.
Change in Self-Rated Health Measured by Visual Analogue Scale (EQ-VAS) | Baseline, 6 months, and 12 months after first MUSE cell treatment
  Self-perceived overall health status will be assessed using the EuroQol Visual Analogue Scale (EQ-VAS). The EQ-VAS is a validated vertical visual analogue scale on which participants rate their current health status. Scale range: 0 to 100
  0 = Worst imaginable health state
  100 = Best imaginable health state
  Interpretation: Higher EQ-VAS scores indicate better self-rated health
  Changes in EQ-VAS scores will be evaluated from baseline to follow-up assessments.
  Proxy-reported responses will be permitted when participants are unable to self-report due to neurological impairment.
Change in Tumor Necrosis Factor Alpha (TNF-α) Serum Concentration | Baseline, 3 months, and 6 months after first MUSE cell treatment
  Serum concentrations of Tumor Necrosis Factor Alpha (TNF-α), a pro-inflammatory cytokine implicated in neuroinflammation and secondary injury following traumatic brain injury, will be obtained when available from participants' independently ordered clinical laboratory tests. TNF-α values will be abstracted from medical records or participant-provided laboratory reports. No laboratory testing or biospecimen collection is performed by the study team.
  Unit of measure: picograms per milliliter (pg/mL)
  Interpretation: Higher TNF-α concentrations indicate greater inflammatory activity
  Changes in TNF-α concentrations will be evaluated between baseline and follow-up time points.
Change in C-Reactive Protein (CRP) Serum Concentration | Time Frame: Baseline, 3 months, and 6 months after first MUSE cell treatment
  Serum concentrations of C-Reactive Protein (CRP), a systemic inflammatory biomarker commonly associated with chronic inflammation and injury response, will be obtained when available from participants' independently ordered clinical laboratory tests. CRP values will be abstracted from medical records or participant-provided laboratory reports. The study does not order laboratory testing or collect biospecimens.
  Unit of measure: milligrams per liter (mg/L)
  Interpretation: Higher CRP concentrations indicate greater systemic inflammation
  Changes in CRP concentrations will be evaluated between baseline and follow-up time points.

OTHER OUTCOMES:
Change in health care utilization related to traumatic brain injury | 12 months before and 12 months after first MUSE cell treatment
  Health care utilization related to traumatic brain injury-including emergency department visits, unplanned hospitalizations, and outpatient neurology or rehabilitation visits-will be abstracted from participant reports and available medical records. This outcome will assess differences in the number of TBI-related visits or hospitalizations per participant-year when comparing the 12 months prior to the participant's first independently obtained MUSE cell therapy session with the 12 months following that session. All data reflect routine medical care and are not influenced or directed by the study.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Lambert Abeyatunge, MD: Regenerative Medicine, Principal Investigator
Locations (2):
- Healing Hope International, Houston, Texas, United States
- Stem Solutions, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Uchida H, Niizuma K, Kushida Y, Wakao S, Tominaga T, Borlongan CV, Dezawa M. Human Muse Cells Reconstruct Neuronal Circuitry in Subacute Lacunar Stroke Model. Stroke. 2017 Feb;48(2):428-435. doi: 10.1161/STROKEAHA.116.014950. Epub 2016 Dec 20. PMID 27999136
- [Background] Abe T, Aburakawa D, Niizuma K, Iwabuchi N, Kajitani T, Wakao S, Kushida Y, Dezawa M, Borlongan CV, Tominaga T. Intravenously Transplanted Human Multilineage-Differentiating Stress-Enduring Cells Afford Brain Repair in a Mouse Lacunar Stroke Model. Stroke. 2020 Feb;51(2):601-611. doi: 10.1161/STROKEAHA.119.026589. Epub 2019 Dec 12. PMID 31826733
- [Background] Yamauchi T, Kuroda Y, Morita T, Shichinohe H, Houkin K, Dezawa M, Kuroda S. Therapeutic effects of human multilineage-differentiating stress enduring (MUSE) cell transplantation into infarct brain of mice. PLoS One. 2015 Mar 6;10(3):e0116009. doi: 10.1371/journal.pone.0116009. eCollection 2015. PMID 25747577
- See also: Related Info — https://www.musestemcelltherapy.com